CLINICAL TRIAL: NCT06496022
Title: Comparative Analysis of Risk Factors and Prediction of Frailty Syndrome
Acronym: FRAILTY-KZ
Status: Active, not recruiting | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Indira Omarova, Principal Investigator, Assistant of the department of General Medical Practice, Asfendiyarov Kazakh National Medical University
Other Study IDs: 01-050124
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Frail Elderly Syndrome
Keywords: frailty; elderly; risk factors; prediction
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort: Patients will be divided into 2 groups: pre-frailty and frailty using Frail Scale.
  Interventions: Diagnostic Test: Frail scale; Diagnostic Test: Barthel scale; Diagnostic Test: SARC-F; Diagnostic Test: FRAX; Diagnostic Test: Mini-Cog scale; Diagnostic Test: dynamometry

INTERVENTIONS:
Diagnostic Test: Frail scale — FRAIL scale for determining frailty (tired most of the time in the last 4 weeks; the presence of more than 5 diseases; difficulty or inability when climbing stairs and walking around the block; weight loss of more than 5% of the previous weight in the last 6 months).
Diagnostic Test: Barthel scale — The Barthel scale is used to determine the degree of independence in daily life, the patient's household activity, the assessment of the quality of life and the necessary care.
Diagnostic Test: SARC-F — The SARC-F scale is used to identify muscle dysfunction (difficulty lifting things over 4.5 kg, walking around the room, difficulty climbing from a chair and up 10 steps, whether the respondent has fallen in the last year).
Diagnostic Test: FRAX — FRAX Scale (Kazakhstan platform) fracture and osteoporosis risk assessment on the website https://frax.shef.ac.uk/FRAX/tool.aspx?country=72
Diagnostic Test: Mini-Cog scale — The Mini-Cog scale defines cognitive impairment (cognitive impairment - when scoring less than 3 points based on remembering three words and evaluating the task of drawing a clock).
Diagnostic Test: dynamometry — carpal dynamometry (sarcopenia is exhibited at values below 26 units for men and below 16 units for women).

SUMMARY:
Assessing frailty syndrome in elderly patients in Almaty To study the features of the clinical course in the group of patients with a pre-frailty and in the group with frailty syndrome

DETAILED DESCRIPTION:
2 cohorts of patients: a group of patients with pre-frailty (300 patients) and a group of patients with frailty syndrome (300 patients).

Comparative analysis of the indicators of two groups (demographic, laboratory indicators, scale results).

To study the features of the clinical course of frailty. To determine the risk factors for the development of frailty. To identify criteria for an unfavorable outcome of frailty.

The study will involve patients over the age of 60. The recruitment of patients will be carried out in polyclinics and nursing homes in Kazakhstan.

The collection of primary information and a comprehensive examination of patients will be based on the following research methods recommended by WHO:

1. Measurements of anthropometric data for calculating body mass index.
2. orthostatic test (active) with measurement of blood pressure, heart rate in horizontal and vertical positions. Blood pressure is measured by the auscultative method (Korotkov method).
3. Survey-based tests:

   * the Bartel scale for determining the degree of independence in daily life, the patient's household activity, assessing the quality of life and the necessary care.
   * The Food Frequency Questionnaire on food preferences over the last 4-week period and the MNA questionnaire on the detection of malnutrition
   * FRAIL scale for determining senile asthenia (tired most of the time in the last 4 weeks; presence of more than 5 diseases; difficulty or inability when climbing stairs and walking around the block; weight loss of more than 5% of the previous weight in the last 6 months).
   * SARC-F scale for detecting muscle dysfunction (difficulty lifting things over 4.5 kg, walking around the room, difficulty climbing from a chair and up 10 steps, whether the respondent has fallen in the last year).
   * FRAX scale (Kazakhstan platform) assessment of fracture and osteoporosis risk on the website https://frax.shef.ac.uk/FRAX/tool.aspx?country=72
   * Mini-Cog scale for determining cognitive impairment (cognitive impairment - when scoring less than 3 points based on remembering three words and evaluating the task of drawing a clock).
4. carpal dynamometry (sarcopenia is exhibited at values below 26 units for men and below 16 units for women).
5. Laboratory parameters: uric acid, serum creatinine calculated using the CKD-EPI formula, creatinine clearance according to the Cockcroft-Gault formula, blood iron levels, blood ferritin, vitamin B12 in the blood, folate in the blood, total protein and albumin in the blood, 25-OH vitamin D in the blood.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 60 years of age
2. Signatories of the informed consent to participate in the study

Exclusion Criteria:

1. Not agreeing to participate in scientific research
2. Elderly people who do not understand the purpose of the study
3. Severe and decompensated diseases that do not allow the study.
4. Concomitant oncological diseases
5. Concomitant neurological and mental disorders that impede the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients from polyclinics of nursing homes in Kazakhstan
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
frailty prevalence | 1 March 2024 - 31 December 2024
  A FRAIL scale or Fried frailty criteria is used (weight loss, exhaustion, low physical activity, slowness, weakness). The participants were divided into three stages: non-frail (score 0), pre-frail (score 1-2) and frail (score 3-5).

CONTACTS AND LOCATIONS:
Locations (1):
- Kazakh National Medical University, Almaty, Tole Bi 94, Kazakhstan

IPD SHARING:
Plan to Share IPD: No
patients data is available upon request from the authors with no identifiable information